CLINICAL TRIAL: NCT05056766
Title: How Does the Clinical and Paraclinical Efficacy of an Oral Appliance Evolve According to Propulsion: Control With Each mm of Advancement"
Brief Title: How Does the Clinical and Paraclinical Efficacy of an Oral Appliance Evolved According to Propulsion: Control With Each mm of Advancement
Acronym: OAMMM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-03
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiratory Tract Diseases
Keywords: oral appliance
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group assignement
  Interventions: Behavioral: questionnaires: Epworth Sleepiness Scale; Pichot fatigue questionnaire.

INTERVENTIONS:
Behavioral: questionnaires: Epworth Sleepiness Scale; Pichot fatigue questionnaire. — Each patient will undergo 3 to 7 polygraphy recordings according usual practice of titration At the same time, Self-questionnaires will be conducted by the patient in order to evaluate Oral appliance efficacy.
  Optimal titration of oral appliance will be done according subjectives parameters. (sleepeness Reduction and fatigue Reduction).
  Neither the investigator nor the patient will know the polygraphy results (apnea-hypopnea index)

SUMMARY:
The OAMMM study is a mono-centrer , non interventional, prospective study, carried out in CH Valence

Oral Appliance is indicated for first line moderate sleep Apnea Syndrome or severe sleep Apnea Syndrome after failure of positive airway pressure (CPAP).

Clinical impact of each mm advancement of Oral Appliance is imperfectly assessed.

The study aim to assess clinical and paraclinical efficacy of an oral Appliance on each mm of advancement.

DETAILED DESCRIPTION:
Oral appliance will be delivered with a propulsion at 50% of the maximum advance and the investigator will titrate the advance according to the usual method

Polygraphy and clinical effectiveness of the Oral appliance will be evaluate

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Moderate sleep apnea diagnosis with clinical signs
* Severe sleep apnea with failure continuous positive airway pressure( CPAP)

Exclusion Criteria:

* previous sleep apnea treatment for Moderate sleep apnea
* refusal to participate in research
* Patient under guardianship, deprived of liberty, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients, with primary Moderate sleep apnea or Severe sleep apnea with failure continuous positive airway pressure( CPAP).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 6 months
  severity of sleep apnea

SECONDARY OUTCOMES:
Epworth Sleepiness Scale score | 6 months
pichot fatigue questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BUIRET, MD, Principal Investigator — CH VALENCE
Locations (1):
- CH Valence, Valence, France